CLINICAL TRIAL: NCT01494883
Title: Mindfulness Based Stress Reduction (MBSR) for Patients With Lung Cancer and Their Partners: a Randomized Controlled Trial.
Brief Title: Mindfulness for Lung Cancer Patients and Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MFN 2011-2015
Record Dates: First submitted 2011-12-02; First posted 2011-12-19 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Lung Cancer
Keywords: Mindfulness Based Stress Reduction; lung cancer; psychological distress; caretakers
MeSH Terms: conditions — Lung Neoplasms | interventions — Mindfulness-Based Stress Reduction

ARMS (2):
- Treatment as usual (No Intervention)
- Mindfulnes Based Stress Reduction (Experimental): A weekly training of eight session lasting two and a half hours.
  Interventions: Behavioral: Mindfulness Based Stress Reduction

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — A weekly training of eight sessions lasting two and a half hours.
  Arms: Mindfulnes Based Stress Reduction

SUMMARY:
The aim of the current study is to examine the (cost)effectiveness of mindfulness based stress reduction (MBSR) in comparison with treatment as usual for patients with lung cancer and their partners.

DETAILED DESCRIPTION:
Receiving a diagnosis of cancer is a major cause of distress and is usually characterized by anxiety and depression. Compared to patients with other cancer diagnoses, patients with lung cancer report higher levels of distress, which probably can be explained by the poor prognosis. At the time of diagnosis, lung cancer is often locally or systematically advanced and 5-year survival is only 15 percent.

Mindfulness based stress reduction (MBSR) is a recently developed psychological intervention that appears to be promising in terms of reducing psychological distress in cancer patients. It consists of 8 weekly group sessions in which formal and informal mindfulness practices are practiced. As most of the earlier studies have been conducted in patients with breast cancer, it is important to examine the effectiveness of this approach in patients with other types of cancer, such as lung cancer. Furthermore, a diagnosis of cancer is not only highly distressing for the patient but also for the partner and family.

In this study, the (cost)effectiveness of MBSR compared with treatment as usual will be investigated in 110 patients with lung cancer and 110 partners.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically proven non-small cell lung cancer and small cell lung cancer.
* Patients can participate after lung cancer diagnosis, from start of treatment or after treatment.
* Sufficient understanding of Dutch language.

Exclusion Criteria:

* Former participation in MBSR or MBCT course.
* Current psychological treatment by psychologist or psychiatrist.
* Cognitive impairments hampering participation in MBSR and completion of questionnaires.
* Physical impairments prohibiting participation in MBSR training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Psychological Distress at 3 and 6 months | at 0, 3, 6 months

SECONDARY OUTCOMES:
Change from baseline in Marital satisfaction at 3 and 6 months | at 0, 3, 6 months
Change from baseline in Quality of Life at 3 and 6 months | at 0, 3, 6 months
Change from baseline in Medical costs at 3 and 6 months | at 0, 3, 6 months
Change from baseline in Mindfulness Skills at 3 and 6 months | 0, 3, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne EM Speckens, Prof. dr., Principal Investigator — Radboud University Medical Center; Miep A van der Drift, Drs., Principal Investigator — Radboud University Medical Center; Judith B Prins, Prof. dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre for Mindfulness, Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Schellekens MP, van den Hurk DG, Prins JB, Molema J, Donders AR, Woertman WH, van der Drift MA, Speckens AE. Study protocol of a randomized controlled trial comparing Mindfulness-Based Stress Reduction with treatment as usual in reducing psychological distress in patients with lung cancer and their partners: the MILON study. BMC Cancer. 2014 Jan 3;14:3. doi: 10.1186/1471-2407-14-3. PMID 24386906